CLINICAL TRIAL: NCT04783584
Title: Agreement Between Video and In-person Airway Assessment Performed by Anaesthetists in Patients Scheduled for Elective Same-day Gynaecological Procedures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Michael Ma (Other)
Responsible Party: Sponsor-Investigator, Michael Ma, Locum Consultant, Coombe Women and Infants University Hospital
Organization: Coombe Women and Infants University Hospital (Other)
Other Study IDs: Study No. 25 - 2020
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Difficult Intubation; Difficult Airway Intubation
Keywords: Pre-operative airway assessment; Virtual airway assessment; Airway examination; Pre-operative airway examination; Airway Tests; Difficult airway prediction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During a general anaesthetic, patients cannot breathe on their own and have to be artificially ventilated. This is achieved by connecting the patient's windpipe (trachea) to a ventilator via the use of a plastic tube called an endotracheal tube (ETT). To place this ETT into the patient's trachea, an instrument called a laryngoscope is used to lift the tongue and view the entrance to the trachea. This process is called laryngoscopy. The act of placing this ETT into the trachea is called intubation.

In anticipation of this procedure, the airway is assessed by the anaesthetist before the patient is put to sleep. This airway examination helps predict if the patient's airway will prove to be difficult to intubate. This assessment is usually carried out face to face with the patient.

Since the onset of the COVID 19 pandemic, we have been trying to minimise patient footfall performing anaesthetic assessments before surgery through a video platform. The objective of this study is to compare these video airway evaluations to assessments carried out face to face.

We anticipate that the virtual airway assessments will be similar if not the same as the in-person airway assessments.

DETAILED DESCRIPTION:
This is a prospective observational study. We are comparing the agreement between a virtual video airway evaluation and an inpatient person-to-doctor airway assessment.

Patients will be referred for virtual preoperative assessment clinic by the gynaecology outpatient department based on inclusion criteria and a patient information leaflet and consent form is supplied at this time. During the virtual assessment consent is taken, followed by a standard history and airway examination. The airway assessment will be performed by an investigator of >5 years anaesthetic experience and will have to undergo a standardised airway assessment training. This airway evaluation is also documented separate to the remainder of the history, sealed in an envelope and labelled a designated number. On the date of surgery, the patient is assessed again by an investigator in the ward/theatre prior to surgery. This airway examination is documented on the standard anaesthetic record sheet as well as on a separate in-person evaluation form. This airway assessment form is then sealed in an envelope and labelled the same designated number as the virtual assessment. The evaluations will be entered into a database and analysed.

If the evaluation is found to show predictors of a difficult airway in the virtual clinic, the patient is scheduled for an in-person outpatient appointment. The airway is then assessed by an investigator in-person at the clinic. The airway is then assessed by an anaesthetic consultant and documented on the anaesthetic record sheet. Investigators will have no further involvement in the clinical management of the patient.

ELIGIBILITY:
Inclusion Criteria:

* We will include patients attending clinic for minor or intermediate gynaecological surgery who were ASA physical status 1-2, BMI less than 40, greater than 18 and less than 65 years of age and no language barrier.

Exclusion Criteria:

* We excluded anyone over 65 years of age, with a BMI over 40, ASA physical status over 2, undergoing major gynaecological surgery, requiring translation services or difficulty accessing virtual technology.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — The study includes patients going for gynaecological procedures and as such only pertains to the female gender
Study Population: The population is from patients attending clinic for minor or intermediate gynaecological surgery in the Coombe Women & Infants University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Agreement between virtual and in-person airway examinations | 6 months
  To determine whether the airway assessment via a virtual platform is in agreement with an in-person airway examination in patients scheduled for elective day-surgery procedures.

SECONDARY OUTCOMES:
Agreement between virtual and in-person airway assessments in suspecting a difficult airway | 6 months
  To compare the overall airway evaluation between clinicians using the video platform versus in-person assessments as binary outcome - difficult airway suspected or not suspected.

CONTACTS AND LOCATIONS:
Locations (1):
- The Coombe Women & Infants University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided